CLINICAL TRIAL: NCT03751410
Title: Long-term Effect of Chronic Ibrutinib Therapy on Left Atrial Function
Brief Title: Chronic Ibrutinib Therapy Effect on Left Atrial Function
Acronym: CITE-LA
Status: Completed | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Ivan Zeljkovic, Principal co-investigator, University Hospital Sestre Milosrdnice
Other Study IDs: UHS-2; U1111-1221-9732 (Other: Universal Trial Number - World Health Organization)
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Atrium; Beat; Echocardiography; Physiology; Therapy Adverse Effect
Keywords: ibrutinib; echocardiography; left atrium; function; long-term

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ibrutinib is an irreversible Bruton tyrosine-kinase inhibitor. In prospective studies, the ibrutinib efficacy in the treatment of various B-cell malignancies was established. Different ibrutinib side-effects have been found: diarrhea, arthralgia, infections, neutropenia, hypertension and increased risk of bleeding. Most of the mentioned side-effects were <3rd degree of severity and mostly didn't require dose adjustment or therapy discontinuation. Also, there was an increase in the incidence of atrial fibrillation (AFib) (6-16%). The AFib pathogenesis in this patient population is not clarified, but there are indications that ibrutinib inhibits phosphoinositide-3-kinase (PI3K)-Akt signal-pathway expressed in the myocytes. Regardless of the molecular pathogenesis, the clinical effect of ibrutinib on the myocardium, especially the left atrium, has not been studied. Hence, the aim of this study is to determine the ibrutinib effect on echocardiographic parameters of left atrial function.

This study will be performed as a clinical, prospective, observational cohort study with a structured follow-up period of 12 months. All consecutive patients with hemato-oncologic diseases (including chronic lymphocytic leukemia, Mantle-cell lymphoma, Waldenstrom macroglobulinemia, etc.) prescribed with chronic ibrutinib therapy, who are able to understand and sign informed consent, will be enrolled. Primary objective is change of the left atrial function measured by the decrease of the left atrial strain deformation > 10%.

Recruiting should not exceed 12 months with the minimal follow-up period of 12 months (24 months in total). Standardized statistical methods and tests will be done using SPSS Version 22.0 or newer.

This unique study offers the possibility to show the long-term effect of chronic ibrutinib therapy on left atrial function assessed by transthoracic echocardiography. This observational data is needed to further refine the treatment of these patients and to prevent possible side-effects of ibrutinib which could endanger this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* patients with haemato-oncologic diseases (including chronic lymphocytic leukemia, Mantle-cell lymphoma, Waldenstrom macroglobulinaemia, etc.)
* patients prescribed with chronic ibrutinib therapy
* patients who are able to understand and sign informed consent

Exclusion Criteria:

* patients with haemato-oncologic diseases who were prescribed with concomitant chemotherapy which can impact left atrial function
* patients < 18 years old
* patients with known or at initial echocardiography established dilated cardiomyopathy with left ventricular ejection fraction < 35%
* patients with permanent atrial fibrillation and dilated left atrium or dilated both atriums
* patients implanted with cardiac implantable electronic devices
* patients who underwent cardiac surgery
* patients with congenital heart diseases (surgically corrected or not)
* patients with severe valvular pathology
* patients with terminal renal disease
* patients with chronic obstructive pulmonary disease - GOLD grade 4
* patients with life expectancy < 12 months
* patients not willing to undergo clinical follow-up or sign informed consent
* patients recruited in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with haemato-oncologic diseases (including chronic lymphocytic leukemia, Mantle-cell lymphoma, Waldenstrom macroglobulinaemia) prescribed with chronic ibrutinib therapy, who are able to understand and sign informed consent, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
left atrial function change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  change of the left atrial function measured by the decrease of the left atrial strain deformation > 10% assessed by transthoracic echocardiography

SECONDARY OUTCOMES:
left ventricular ejection fraction change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  measurement of left ventricular systolic function change assessed by transthoracic echocardiography - method according to Simpson and Teicholz
left ventricular diastolic function change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  measurement of left ventricular diastolic function change assessed by transthoracic echocardiography (E/A and E/E')
left atrial volume change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  2D and 3D left atrial volume change assessed by transthoracic echocardiography + left atrial dimension in PLAX and 4 chamber projection
P wave duration change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  P wave duration and PQ interval duration change assessed in 12-lead electrocardiogram (in milliseconds)
left atrial pump function change | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  left atrial ejection fractionchange assessed by transthoracic echocardiography (doppler strain measurement method)
atrial fibrillation incidence | initial measurement, 3 months, 6 months and 12 months after initiation of ibrutinib therapy
  incidence of paroxysmal atrial fibrillation assessed by symptoms + ECG or 24-hours Holter-ECG

CONTACTS AND LOCATIONS:
Overall Officials: Matea Kolacevic, MD, Principal Investigator — University Hospital Sestre Milosrdnice
Locations (1):
- Sestre milosrdnice University Hospital, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deeks ED. Ibrutinib: A Review in Chronic Lymphocytic Leukaemia. Drugs. 2017 Feb;77(2):225-236. doi: 10.1007/s40265-017-0695-3. PMID 28105602
- [Result] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Result] Thompson PA, Burger JA. Bruton's tyrosine kinase inhibitors: first and second generation agents for patients with Chronic Lymphocytic Leukemia (CLL). Expert Opin Investig Drugs. 2018 Jan;27(1):31-42. doi: 10.1080/13543784.2018.1404027. Epub 2017 Nov 15. PMID 29125406
- [Result] Wierda WG, Zelenetz AD, Gordon LI, Abramson JS, Advani RH, Andreadis CB, Bartlett N, Byrd JC, Caimi P, Fayad LE, Fisher RI, Glenn MJ, Habermann TM, Harris NL, Hernandez-Ilizaliturri F, Hoppe RT, Horwitz SM, Kaminski MS, Kelsey CR, Kim YH, Krivacic S, LaCasce AS, Martin MG, Nademanee A, Porcu P, Press O, Rabinovitch R, Reddy N, Reid E, Roberts K, Saad AA, Snyder ED, Sokol L, Swinnen LJ, Vose JM, Yahalom J, Dwyer MA, Sundar H. NCCN Guidelines Insights: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma, Version 1.2017. J Natl Compr Canc Netw. 2017 Mar;15(3):293-311. doi: 10.6004/jnccn.2017.0030. PMID 28275031
- [Result] Burger JA, Tedeschi A, Barr PM, Robak T, Owen C, Ghia P, Bairey O, Hillmen P, Bartlett NL, Li J, Simpson D, Grosicki S, Devereux S, McCarthy H, Coutre S, Quach H, Gaidano G, Maslyak Z, Stevens DA, Janssens A, Offner F, Mayer J, O'Dwyer M, Hellmann A, Schuh A, Siddiqi T, Polliack A, Tam CS, Suri D, Cheng M, Clow F, Styles L, James DF, Kipps TJ; RESONATE-2 Investigators. Ibrutinib as Initial Therapy for Patients with Chronic Lymphocytic Leukemia. N Engl J Med. 2015 Dec 17;373(25):2425-37. doi: 10.1056/NEJMoa1509388. Epub 2015 Dec 6. PMID 26639149
- [Result] Kaur V, Swami A. Ibrutinib in CLL: a focus on adverse events, resistance, and novel approaches beyond ibrutinib. Ann Hematol. 2017 Jul;96(7):1175-1184. doi: 10.1007/s00277-017-2973-2. Epub 2017 Mar 24. PMID 28342031
- [Result] O'Brien S, Hillmen P, Coutre S, Barr PM, Fraser G, Tedeschi A, Burger JA, Dilhuydy MS, Hess G, Moreno C, Cramer P, Liu E, Chang S, Vermeulen J, Styles L, Howes A, James DF, Patel K, Graef T, Valentino R. Safety Analysis of Four Randomized Controlled Studies of Ibrutinib in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Mantle Cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2018 Oct;18(10):648-657.e15. doi: 10.1016/j.clml.2018.06.016. Epub 2018 Jun 28. PMID 30061088
- [Result] Reda G, Fattizzo B, Cassin R, Mattiello V, Tonella T, Giannarelli D, Massari F, Cortelezzi A. Predictors of atrial fibrillation in ibrutinib-treated CLL patients: a prospective study. J Hematol Oncol. 2018 Jun 11;11(1):79. doi: 10.1186/s13045-018-0626-0. PMID 29891001
- [Result] Boriani G, Corradini P, Cuneo A, Falanga A, Foa R, Gaidano G, Ghia PP, Martelli M, Marasca R, Massaia M, Mauro FR, Minotti G, Molica S, Montillo M, Pinto A, Tedeschi A, Vitolo U, Zinzani PL. Practical management of ibrutinib in the real life: Focus on atrial fibrillation and bleeding. Hematol Oncol. 2018 Oct;36(4):624-632. doi: 10.1002/hon.2503. Epub 2018 Mar 7. PMID 29512173
- [Result] Mato AR, Clasen S, Pickens P, Gashonia L, Rhodes J, Svoboda J, Hughes M, Nabhan C, Ali N, Schuster S, Carver J. Left atrial abnormality (LAA) as a predictor of ibrutinib-associated atrial fibrillation in patients with chronic lymphocytic leukemia. Cancer Biol Ther. 2018 Jan 2;19(1):1-2. doi: 10.1080/15384047.2017.1394554. Epub 2017 Dec 27. PMID 29281559
- [Result] Leong DP, Caron F, Hillis C, Duan A, Healey JS, Fraser G, Siegal D. The risk of atrial fibrillation with ibrutinib use: a systematic review and meta-analysis. Blood. 2016 Jul 7;128(1):138-40. doi: 10.1182/blood-2016-05-712828. Epub 2016 May 31. No abstract available. PMID 27247135